CLINICAL TRIAL: NCT00872196
Title: A Follow-up Study to Assess the Evolution and Persistence of Resistance to ABT-072 After Discontinuation of ABT-072 Therapy in HCV Genotype-1 Infected Subjects Who Participated in Phase 1, 2, or 3 ABT-072 Clinical Studies
Brief Title: A Follow-up Study to Assess Resistance to ABT-072 in HCV-infected Subjects Administered ABT-072 in Prior ABT-072 Studies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M10-605
Record Dates: First submitted 2009-03-23; First posted 2009-03-31 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — ABT-072

ARMS (1):
- 1 - Follow-up Study (Other): This is a follow-up study with no treatment and only samples being collected.
  Interventions: Drug: ABT-072

INTERVENTIONS:
Drug: ABT-072 — Blood samples are being taken from subjects previously treated with ABT-072.

SUMMARY:
This is a follow-up study with no treatment and only samples being collected.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the development of specific viral mutations in response to treatment with ABT-072.

ELIGIBILITY:
Inclusion Criteria:

- Main Selection Criteria: A subject that has received either ABT-072 or placebo in a prior study involving ABT-072.

Exclusion Criteria:

- The investigator considers the subject unsuitable for the study for any reasons inclusive of, but not limited to, failure to comply with study procedures in a prior ABT-072 clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Analysis of the prevalence of resistance of specific mutations over time will be summarized. | Approximately 48 weeks.
Analysis of the degree of phenotypic resistance (fold change in susceptibility of ABT-072 compared to wild-type virus) will also be summarized. | Approximately 48 weeks.

SECONDARY OUTCOMES:
Summary of serious adverse events related to study procedures only. | Approximately 48 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — AbbVie
Locations (1):
- Site Reference ID/Investigator# 18222, Los Angeles, California, United States